CLINICAL TRIAL: NCT04881500
Title: Impact of a Brief Motivational Intervention Including Counter-marketing Arguments With a Population of Patients With Moderate to Severe Alcohol Use Disorders Who Are Followed up on an Outpatient Basis (Primary Care or Addictology)
Brief Title: Impact of a Brief Motivational Intervention Including Counter-marketing Arguments With a Population of Patients With Moderate to Severe Alcohol Use Disorders Who Are Followed up on an Outpatient Basis (Primary Care or Addictology) (DEPREV_Phase 3)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting difficulties
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC20.0261
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Addiction, Alcohol
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interview (Experimental): Patients followed in the primary care network participating in the study and those followed in the addictology network of northern Finistère in the context of their pathology will be offered the opportunity to participate in the study.
  If the patient was randomized to the intervention group, the patient will receive 2 individual sessions (motivational interview) by telephone within 1 month of inclusion. They will then be assessed at month 1, month 3 and month 6. These assessments will be done by telephone.
  Interventions: Other: Motivational interview
- Routine Care (Active Comparator): Patients followed in the primary care network participating in the study and those followed in the addictology network of northern Finistère in the context of their pathology will be offered the opportunity to participate in the study.
  If the patient has been randomized to the control group, the patient will be assessed at month 1, month 3 and month 6. These assessments will be done by telephone.
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Motivational interview — Patients will follow motivational interview (2 individual sessions by phone)
  Arms: Motivational interview
Other: Routine Care — Patients will follow routine care
  Arms: Routine Care

SUMMARY:
Alcohol consumption is the second cause of avoidable death after tobacco. The Evin law was constructed in 1991 with the aim of reducing exposure to alcohol marketing among the youngest. But this law is currently extremely weakened, and in a press release of February 26, 2018, the French Alcohol Society is alarmed by these developments.

Studies on the impact of alcohol marketing focus for the most part on young adolescents and the links between marketing exposure and alcohol initiation. But beyond these links, little work has been done on the impact of alcohol marketing on vulnerable subjects with regular alcohol consumption. Alcohol consumption is one of the very first causes of hospitalization in France. The damage is often limited to the notion of risks of dependence, but it can appear as soon as consumption of 1 standard unit/day and mainly concerns the 45-64 year olds. To our knowledge, there are no studies on the impact of alcohol marketing carried out among regular alcohol users with moderate or severe alcohol use disorders. This population is, however, the target of manufacturers, since 10% of the French population consumes 58% of the alcohol sold in France. Moreover, although in the context of tobacco, counter-marketing campaigns and strategies are used to help users develop resistance to the positive marketing stimuli of alcohol, there are no studies that have evaluated this type of intervention with patients with moderate to severe alcohol use disorders.

The DEPREV_phase 3 study is a prospective, controlled, randomised, open-label study.

Patients followed in the primary care network participating in the study and those followed in the addictology network of northern Finistère in the context of their pathology will be offered the opportunity to participate in the study.

Patients agreeing to participate will be randomized in 2 groups (1:1) by the addictology unit:

* Control group: routine routine follow-up (follow-up in consultations with the attending physician or addictologist) + assessments at Month 1, Month 3 and Month 6.
* Intervention group: Routine routine follow-up (follow-up in consultation with the attending physician or addictologist) + assessments at Month 1, Month 3 and Month 6 + motivational interview (2 individual sessions, during the first month after inclusion).

Patients will then be followed up and evaluated at 1, 3 and 6 months after the inclusion visit.

ELIGIBILITY:
Inclusion Criteria :

- Patient over 18 years of age

* Current alcohol consumption (several times a month)
* Compliance with the criteria for harmful use or dependence according to AUDIT scale greater than or equal to 7 for men or 6 for women
* Outpatient follow-up in primary care or in addictology in the addictology network of northern Finistère

Exclusion Criteria :

* Patient under 18 years of age
* Subject under legal protection, guardianship, or curatorship or deprived of liberty
* Non comprehension of the French language
* Acute unstable psychiatric disorders affecting judgment
* No fixed or cell phone line
* AUDIT score less than 6 for women and 7 for men
* Addictology hospitalization history in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Ability of patients to control their own alcohol consumption | Day 0 to Month 6
  The primary outcome is the perceived ability of patients to control their own alcohol consumption measured on a visual analogue scale from 0 to 100 in relation to the question "How much do you estimate your ability to control your alcohol consumption?" with 0 = no ability to control my drinking and 100 = all my ability to control my drinking. This primary outcome is evaluated at 3 month.

SECONDARY OUTCOMES:
Evaluation of quality of life | Day 0, Month 1, Month 3 and Month 6
  The quality of life will be evaluated by AQoLS scale whose is a specific quality of life scale to alcohol use disorders. It measures the negative impact of the relationship with alcohol on quality of life through 7 dimensions (Relationships with others, Activities, Negative emotions, Self-esteem, Loss of control, Sleep, Living conditions). Each item corresponds to a score from 0 (not at all) to 3 (very much), the total score being the sum of the 34 items in this self-questionnaire. There is no threshold value, as the patient is his or her own control in his or her own evolution.
Severity of alcohol use disorders | Day 0, Month 1, Month 3 and Month 6
  Severity of alcohol use disorders at each visit, as measured by the AUDIT ( (Alcohol Use Disorders Identification Test) score.
  AUDIT (Alcohol Use Disorders Identification Test) score is a 10-item screening tool to assess alcohol consumption, drinking behaviors, and alcohol-related problems. A score of 8 or more is considered to indicate hazardous or harmful alcohol use.
Evaluation of severity of alcohol use disorders | Day 0, Month 1, Month 3 and Month 6
  Severity of alcohol use disorders at each visit, as measured by the number of DSM5 (Diagnostic and Statistical manual of Mental disorders 5) criteria. The DSM5 score is diagnosis of addiction is based on well-defined criteria set out in the Diagnostic and Statistical manual of Mental disorders (DSM), the fifth edition of which was published in 2013. The questionnaire consists of 11 items (diagnostic criteria for substance use disorders from the American Psychiatric Association's DSM V). The presence of 2 to 3 criteria: low addiction / Presence of 4 to 5 criteria: moderate addiction / Presence of 6 or more criteria: severe addiction.
Limitation of alcohol consumption | Day 0, Month 1, Month 3 and Month 6
  Ability to implement limiting strategies, as measured by the visual analogue scale from 0 to 100 on the question "How well do you feel you are able to implement strategies to limit/restrict (or avoid) your alcohol consumption" at each visit?
Evaluation of alcohol use | Day 0, Month 1, Month 3 and Month 6
  Alcohol consumption measured by the Alcohol Timeline Followback (ATLFB) score at each visit. The ATLFB (Alcohol Timeline FollowBack) is a method for assessing recent drinking behavior. It involves asking clients to retrospectively estimate their daily alcohol consumption over a time period for 30 days prior to the interview. This scale is just an estimate of alcohol consumption on 1 month, there are no minimum or maximum values and so no better or worse outcome.
Craving assessment | Day 0, Month 1, Month 3 and Month 6
  The Obsessive Compulsive Drinking Scale (OCDS) is a 14-item questionnaire that measures an individual's alcohol use and his/her attempts to control his/her drinking (each item is scored on a scale from 0 to 4). Obsessive subscale is the summation of items 1-6 / Compulsive subscale is the summation of items 7-14.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Guillou Landreat, Brest
  - SIMSON Jean-Pierre, Brest
  - LE GOFF Delphine, Landerneau
  - ROZEC Pascale, Landerneau
  - LE RESTE Jean-Yves, Lanmeur
  - BARAIS Marie, Lannilis

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 19 month and ending 15 years following the final study report completion.
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.